CLINICAL TRIAL: NCT04965519
Title: An Open, Multi-cohort, Multi-center Phase II Basket Clinical Study of RC48-ADC Monotherapy in the Treatment of HER2-expressing (HER2-positive and HER2 Low Expression) Gynecological Malignancies
Brief Title: A Study of RC48-ADC for the Treatment of HER2-expressing Gynecological Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C018
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Gynecological Malignancy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Eligible subjects received RC48-ADC treatment after enrollment, at a dose of 2.0 mg/kg, once every 2 weeks (the dosing time window in all cycles is -1 to 2 days), and the administration method is intravenous Drip.
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — 2.0mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the effectiveness and safety of intravenous injection of RC48-ADC in the treatment of HER2 expression (HER2 positive and HER2 low expression) gynecological malignancies.

DETAILED DESCRIPTION:
This study is an open, multi-cohort, multi-center Phase II basket clinical study that included HER2 expression (HER2 positive and HER2 low expression) gynecological malignant tumor subjects. The four cohorts include cervical cancer, ovarian epithelial cancer、 fallopian tube cancer and primary peritoneal cancer, endometrial cancer and other gynecological malignancies (vulvar cancer, vaginal cancer, primary sarcoma of the gynecological reproductive system, etc.). Each cohort enrolled 30 subjects. Among them, IHC+, IHC2+, IHC3+ subjects were enrolled at least 5 subjects, and the remaining 15 subjects were not restricted by HER2 expression. HER2 expression includes HER2 positive and HER2 low expression. HER2 positive is defined by the immunohistochemical IHC 2+/fluorescence in situ hybridization technique FISH+ or IHC 3+ judged by the central laboratory. HER2 low expression is defined as IHC 2+/FISH- or IHC+ as determined by the central laboratory. The Molecular Pathology Department of the Department of Pathology, Cancer Hospital of the Chinese Academy of Medical Sciences will serve as the research center laboratory to confirm the HER2 status (including IHC and FISH tests).

ELIGIBILITY:
Inclusion Criteria:

* 1. Meet all the conditions of any of the following queues:
* Queue one:

  1. Histologically confirmed patients with recurrent or metastatic cervical cancer who have failed at least the first-line platinum-containing standard treatment or failed concurrent radiotherapy and chemotherapy;
  2. Not suitable for surgery or radiotherapy.
* Queue two:

  1. Ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer confirmed histologically;
  2. The subject has previously received a standard platinum-containing chemotherapy regimen, and at the same time meets any of the following criteria:

Platinum-resistant relapsed patients who have undergone at least 2 lines (can contain BRCA mutations or HRD-positive patients who have failed PARP inhibitors) standard treatment failure (relapse or progression time and previous platinum-containing regimen last chemotherapy (at least 4 cycles) The interval between time is less than 6 months); or at least three lines (patients who have failed PARP inhibitors on BRCA mutations or HRD-positive patients) platinum-sensitive relapsed patients who have failed standard treatment (the time to relapse or progression is related to The interval between the last platinum-containing chemotherapy (at least 4 cycles) is ≥ 6 months); Note: The definition of recurrence or progression (meet any of the following conditions): a) There is clearly recorded imaging progress; b) CA-125 continues to rise (CA-125 ≥ 2 times the upper limit of normal, and it needs to be confirmed after 1 week ) With clinical symptoms or physical examination suggesting disease progression;

* Queue three:

  1. Recurrent or metastatic endometrial cancer confirmed histologically;
  2. Patients who have failed the standard treatment of at least first-line platinum-containing chemotherapy;
  3. Not suitable for surgery or radiotherapy.
* Queue four:

  1. Recurrent or metastatic other gynecological malignancies (vulvar cancer, vaginal cancer, primary sarcoma of the gynecological reproductive system, etc.) that have failed standard treatments confirmed by histology;
  2. Not suitable for surgery or radiotherapy.
* 2.Voluntarily agree to participate in the research and sign an informed consent form;
* 3. Female, age ≥18 years old;
* 4. Expected survival period ≥ 12 weeks;
* 5.The central laboratory confirms the expression of HER2: IHC 1+, 2+ or 3+; the subject can provide specimens of the primary or metastatic tumor site for HER2 detection (paraffin blocks, paraffin-embedded sections or fresh tissue sections are acceptable); IHC2+ Of subjects need to be tested for FISH. Note: The scoring standard for HER2 testing is determined by the central laboratory.
* 6. With measurable lesions specified by RECIST 1.1 standard;
* 7. ECOG physical status 0 or 1 point;
* 8. Sufficient organ functions should meet the following criteria during the screening period (the normal value is subject to the clinical trial center): Left ventricular ejection fraction ≥50%; Hemoglobin ≥9g/dL; Absolute neutrophil count (ANC)≥1.5×109/L; Platelets ≥100 ×109/L; Serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN); ALT and AST≤2.5 × ULN when there is no liver metastasis, and ALT and AST≤5 × ULN when there is liver metastasis; Serum creatinine≤1.5×ULN or calculate creatinine clearance rate (CrCl)≥50 mL/min according to Cockcroft-Gault formula method;
* 9 .Female subjects should be surgically sterilized, post-menopausal patients, or agree to use at least one medically approved contraceptive method (such as intrauterine contraceptive devices, contraceptives, or condom).The blood pregnancy test must be negative within 7 days before study entry, and it must be a non-lactating period.
* 10. Willing and able to follow the trial and follow-up procedures.

Exclusion Criteria:

* 1.Suffering from central nervous system metastasis and/or cancerous meningitis. Subjects who have received brain metastasis therapy may consider participating in this study, provided that the condition is stable for at least 3 months, no disease progression has been confirmed by imaging examination within 4 weeks before the first dose of the study, and all neurological symptoms have recovered At baseline, there is no evidence of new or enlarged brain metastases, and radiation, surgery, or steroid therapy should be discontinued at least 28 days before the first dose of study treatment. This exception does not include cancerous meningitis, which should be excluded regardless of whether the clinical condition is stable or not;
* 2. The toxicity caused by previous anti-tumor treatments has not been restored to CTCAE (version 5.0) 0-1 grade (except for 2nd degree alopecia);
* 3. Major surgery has been performed within 4 weeks before the start of study administration and has not fully recovered;
* 4. A large amount of pleural fluid or ascites accompanied by clinical symptoms or requiring symptomatic treatment;
* 5.Serum virology examination (subject to the normal value of the research center): The HBsAg test result is positive, and the HBV DNA copy number is positive at the same time; HCVAb test result is positive (only if the PCR test result of HCV RNA is negative, it can be selected for this study); HIVAb test result is positive.
* 6. Have received live vaccines within 4 weeks before the start of the study administration or plan to receive any vaccines during the study period (except the new crown vaccination);
* 7. Heart failure classified by the New York College of Cardiology (NYHA) as grade 3 and above;
* 8. Severe arterial/venous thrombotic events or cardiovascular and cerebrovascular accidents occurred within 1 year before the study administration, such as deep vein thrombosis (not including asymptomatic intermuscular vein thrombosis without special treatment), pulmonary embolism, cerebral infarction, Cerebral hemorrhage, myocardial infarction, etc., except for lacunar infarction that is asymptomatic and does not require clinical intervention;
* 9. There are active or advanced infections that require systemic treatment, such as active tuberculosis;
* 10.There are systemic diseases that have not been stably controlled by researchers, including diabetes, hypertension, liver cirrhosis, interstitial pneumonia, obstructive pulmonary disease, etc.;
* 11. There are active autoimmune diseases requiring systemic treatment (such as immunomodulatory drugs, corticosteroids or immunosuppressive agents) within 2 years before the start of study administration, and related alternative treatments (such as thyroxine, insulin, or renal or Physiological corticosteroid replacement therapy for pituitary insufficiency);
* 12. Suffered from other malignant tumors within 5 years before the start of study administration, except for the following conditions: Malignant tumors that can be expected to heal after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ treated by radical surgery);
* 13. Have previously received allogeneic hematopoietic stem cell transplantation;
* 14. Have received other antibody-conjugated drug therapy in the past;
* 15. Those who are known to be allergic to recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent drugs and their components;
* 16. Suffer from any other diseases, metabolic abnormalities, abnormal physical examinations or abnormal laboratory examinations. According to the judgment of the investigator, there is reason to suspect that the patient has a certain disease or condition that is not suitable for the use of the study drug, or will affect the interpretation of the study results , Or put the patient in a high-risk situation;
* 17. It is estimated that the compliance of patients to participate in this clinical study is insufficient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as assessed by the Independent Review Committee | 2 years
  Objective Response Rate is defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Objective Response Rate（ORR）as assessed by investigator | 2 years
  Objective Response Rate is defined as the percentage of participants with a complete response (CR) or partial response (PR)
Duration of Response（DOR） | 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate（DCR） | 2 years
  DCR is defined as the percentage of participants with a complete response (CR), partial response (PR), or stable disease (SD)
Progression Free Survival（PFS） | 2 years
  PFS is defined as the time from the first administration of study treatment to the first occurrence of disease progression or death from any cause, whichever comes first
Overall survival （OS） | 2 years
  OS is defined as the time from the first administration of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality, China